CLINICAL TRIAL: NCT03593694
Title: Technology Delivered Diabetes-Modified Behavioral Activation Treatment for AAs With T2DM
Brief Title: Technology Delivered Diabetes-Modified Behavioral Activation Treatment
Acronym: TECHDMBAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Service provider challenges precluded intervention delivery.
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Ehianu Egede, Professor & Chair, Department of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PRO00030535
Record Dates: First submitted 2018-05-14; First posted 2018-07-20 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Other): Arm: Other: Group 1 Participants in this group will receive the culturally tailored education booklet titled "Your Guide to Sugar Diabetes". In addition, subjects will complete 10 sessions of diabetes education delivered weekly via videoconferencing lasting 60 minutes each session as detailed above.
  Interventions: Behavioral: TECH DMBAT Other
- Group 2 (Active Comparator): Arm: Active Comparator: Group 2 Participants in this group will receive as detailed above, the culturally tailored education booklet titled "My Guide to Sugar Diabetes". In addition, subjects will complete 10 sessions of diabetes education delivered weekly via videoconferencing lasting 60 minutes each session. Patients will also be assigned the FORA Test-n-Go Series Blood Glucose and Blood Pressure monitors and provided glucose test strips to allow testing at least once a day during the initial face-to-face session.
  Interventions: Behavioral: TECH DMBAT Active Comparator
- Group 3 (Experimental): Arm: Experimental: Group 3 The intervention has 3 components: 1) diabetes education; 2) home telemonitoring; and 3) diabetes modified behavioral activation, delivered by nurses via smartphones. Trained nurses will deliver the TECH DM-BAT intervention via videoconferencing technology on smartphones.
  Interventions: Behavioral: TECH DM-BAT

INTERVENTIONS:
Behavioral: TECH DM-BAT — Multi-component, high intensity intervention, technology delivered, diabetes-modified behavioral activation treatment.
  Arms: Group 3
Behavioral: TECH DMBAT Active Comparator — Technology delivered diabetes education and home tele monitoring
  Arms: Group 2
Behavioral: TECH DMBAT Other — Technology delivered diabetes education
  Arms: Group 1

SUMMARY:
The overarching goal of this proposal is to test the efficacy of a multi-component, high intensity intervention, technology delivered, diabetes-modified behavioral activation treatment (TECH DM-BAT) that incorporates: 1) diabetes education; 2) home telemonitoring; and 3) diabetes modified behavioral activation, delivered by nurses via smartphones is effective in improving metabolic control in African Americans with poorly controlled type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes Mellitus is highly prevalent in the United States (CDC 2014) and African Americans (AA) are disproportionately affected and have higher prevalence, poorer metabolic control and greater risk for complications and death compared to White Americans. Evidence from the literature show that effective interventions for AAs with Type 2 Diabetes Mellitus (T2DM) have multiple components including: education and skills training, nurse case management, and maintain high intensity. However, few large Randomized Clinical Trials (RCT) have tested multi-component interventions that include these key components in AAs with T2DM.

Behavioral Activation is a psychotherapeutic process whereby patients are encouraged to identify and schedule structured and enjoyable activities for behavior change that are likely to improve outcomes such as mood, behaviors and quality of life. A brief manualized behavioral activation treatment for depression (BATD), has been modified for diabetes.

This study tests a multi-component, high intensity intervention that incorporates several strategies that have been shown to be effective in improving diabetes outcomes in AAs. Nurse case managers will use videoconferencing technology to deliver education, skills training and problem solving for diabetes via smartphones, an approach that has not been used previously in vulnerable and underserved ethnic minority populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* Clinical diagnosis of T2DM and HbA1c ≥8% at the screening visit;
* Self-identified as AA
* Subject must be willing to use the FORA monitoring system for 6 months
* Subject must be willing to use the study assigned smartphone including videoconferencing, lifestyle monitoring and medication monitoring apps for 6 months
* Subjects must be able to communicate in English
* Subjects must have access to a landline or Ethernet for FORA data uploads for the study period.

Exclusion Criteria:

* Mental confusion on interview suggesting significant dementia
* Participation in other diabetes clinical trials
* Alcohol or drug abuse/dependency
* Active psychosis or acute mental disorder
* Life expectancy <6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Hemoglobin A1c (HbA1c) at 3 and 6 months | baseline, 3-months, 6-months
  Change from Baseline Hemoglobin A1c (HbA1c) at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No